CLINICAL TRIAL: NCT00266734
Title: A Prospective Blinded Multi-center Clinical Trial to Evaluate the Efficacy of the Recently FDA Approved RPS Adeno Detector for Detecting Adenoviral Conjunctivitis
Brief Title: Evaluation of a Rapid Screening Test for Detection of Adenovirus in Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rapid Pathogen Screening (Industry)
Responsible Party: Robert Sambursky, Rapid Pathogen Screening, Inc
Organization: RapidPS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB# 03-543E; St John's IRB# 00003995; Colorado HSC IRB# 05-0151
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Acute Conjunctivitis; Adenoviral Conjunctivitis
Keywords: Adenoviral conjunctivitis; Viral conjunctivitis; conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Viral; Conjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: RPS Adeno Detector

SUMMARY:
To compare the efficacy of a recently FDA approved point of care diagnostic test, the RPS Adeno Detector (Rapid Pathogen Screening, Inc.; South Williamsport, PA), against cell culture for detecting adenoviral conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

Clinical Study Enrollment Criteria

Upon completing the in-vitro studies, a perspective, blinded clinical study was started. Patients who were older than 1 month of age, seen within 7 days of developing a red eye, and who demonstrate at least one criterion from two out of the three categories below were included:

I. History: 1) Spread from one eye to the other several days later, 2) recent or concurrent upper respiratory symptoms within the preceding two weeks, 3) or an exposure to someone with "pink eye" within the preceding three weeks

II. Symptoms: 1) Tearing, 2) mucoid or purulent discharge, 3) eye lash matting, 4) burning, 5) itching, or 6) foreign body sensation

III. Signs: 1) An inferior palpebral conjunctival reaction with > or = 1+ papillary or follicular reactions, 2) presence of a preauricular node

Exclusion Criteria:

Patients with associated skin vesicles, corneal dendrites, traumatic corneal abrasion, concurrent corneal ulcers, foreign bodies, ocular pemphigoid, trauma, previous history of chemical/thermal injury to eyes or eyelids (anytime in past), or greater than trace intraocular inflammation were excluded from the study. Additionally, patients with allergy to corn starch, talcum powder, or dacron were also be excluded. Patients using any topical ophthalmic medication (i.e. antibiotics) were required to wait at least 30 minutes from their last dose prior to device application and wait at least 2 hours after their last dose of any ointment application

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186
Dates: Start 2004-12; Study Completion 2005-09

PRIMARY OUTCOMES:
Ability to accurately detect presence or absence of adenovirus in conjunctival specimens

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth J Cohen, MD, Principal Investigator — Wills Eye Hospital; Shachar Tauber, MD, Principal Investigator — St Johns Ophthalmology Clinic, Springfield, MO; Frank Schirra, MD, Principal Investigator — Universitätsklinikum des Saarlandes, Klinik für Augenheilkunde, Homburg, Germany; Kristian Kozich, MD, Principal Investigator — University of Erlangen-Nurnberg, Erlangen, Germany; Richard Davidson, MD, Principal Investigator — University of Colorado Health Science Center, Denver, CO
Locations (5):
- United States (3):
  - University of Colorado Health Science Center, Denver, Colorado
  - St Johns Ophthalmology Clinic, Springfield, Missouri
  - Wills Eye Hospital, Philadelphia, Pennsylvania
- Germany (2):
  - University of Erlangen-Nurnberg, Erlangen
  - Universitätsklinikum des Saarlandes, Klinik für Augenheilkunde, Homburg